CLINICAL TRIAL: NCT05206890
Title: A Non-interventional Registry Study of Fluzoparib in the Treatment of Ovarian Cancer
Status: Recruiting | Type: Observational
Sponsor: Tongji Hospital (Other)
Collaborators: First Hospital of China Medical University (Other); Cancer Hospital of Xinjiang Medical University (Unknown); First Affiliated Hospital Xi'an Jiaotong University (Other); Qingyuan People's Hospital (Other); Zhejiang University (Other); Panzhihua Central Hospital (Other); Liangshan First People's Hospital (Unknown); Guang'an People's Hospital (Unknown); Afﬁliated Hospital of North Sichuan Medical College (Other); Cancer Hospital of Guizhou Province (Other); Guizhou International General Hospital (Unknown); Yichang Central People's Hospital (Other); Wuhan Fourth Hospital (Unknown); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Qinglei Gao, Professor, Tongji Hospital
Other Study IDs: 2022-TJ-FLU
Record Dates: First submitted 2022-01-11; First posted 2022-01-25 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Ovarian Cancer
Keywords: real world study
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Combined Modality Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — HRD score and BRCA gene test should be conducted using blood and tumor samples. serum CA125 levels should also be tested.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- fluzoparib treatment: patients with Epithelial ovarian cancer, fallopian tube cancer, or primary peritoneal cancer who underwent fluzoparib monotherapy or combination therapy
  Interventions: Drug: fluzoparib monotherapy or combination therapy

INTERVENTIONS:
Drug: fluzoparib monotherapy or combination therapy — patients with epithelial ovarian cancer, fallopian tube cancer or primary peritoneal cancer who underwent fluzoparib monotherapy or combination therapy

SUMMARY:
Ovarian cancer is one of the most fatal malignant tumors that threaten women's health. The incidence rate is the third place among the female reproductive system malignant tumors, and the mortality rate ranks the first in gynecologic malignancies, the majority of patients have advanced diseases at the time of diagnosis.

This observational study is to evaluate the safety and efficacy of fluzoparib in ovarian cancer patients under real conditions, especially in various subgroups of ovarian cancer patients, in order to provide information about treatment modes for ovarian cancer patients in real-world diagnosis and treatment, and preliminarily evaluate the pharmacoeconomic of fluzoparib in the treatment of ovarian cancer.

DETAILED DESCRIPTION:
Ovarian cancer is one of the most serious malignant tumors that threaten women's health. The incidence rate is third place in the female reproductive system malignant tumors. The mortality rate ranks the first in gynecologic malignancies, and most of them are advanced at the time of diagnosis. The initial treatment of ovarian cancer is mainly surgery and adjuvant chemotherapy. Although most patients can obtain clinical remission after initial treatment, 70% of patients still relapse within 3 years. Therefore, finding effective drugs to prolong the chemotherapy-free interval and exploring comprehensive treatment schemes to prolong survival is the key to treatment.

In recent years, the advent of poly adenosine diphosphate ribose polymerase inhibitors has brought significant changes to the treatment of ovarian cancer. A series of high-level evidence-based medical evidence shows that the application of PARP inhibitors after complete and partial remission of initial treatment or platinum-sensitive recurrence treatment can significantly prolong the progression-free survival time of ovarian cancer patients, Maintenance therapy has become a new model for the treatment of ovarian cancer. At the same time, PARP inhibitors have been approved for posterior line treatment of ovarian cancer. At present, PARP inhibitors have been widely used in clinics and become an important cornerstone of the comprehensive treatment of ovarian cancer.

Fzocus-2 study is a multicenter, randomized, double-blind, placebo-controlled phase III clinical study of fluzoparib in the maintenance treatment of platinum-sensitive recurrent ovarian cancer. The preliminary results were published on the American Society of Gynecological Oncology (SGO) in 2021. A total of 252 patients were included in the study and were treated with fluzoparib (n = 167) or placebo (n = 85). The median follow-up time was 8.5 months. The population-wide data assessed by bIRC showed that the median PFS data were not mature. According to the Kaplan Meier curve, fluzoparib could significantly prolong the PFS (12.9 months: 5.5 months) and reduce the risk of disease progression or death by 75%.

Fzocus-3 is a phase IB study of fluzoparib approved for marketing, which included platinum-sensitive recurrent ovarian cancer patients with germline BRCA mutation who had previously received ≥ 3-line treatment. The objective remission rate of single-drug treatment is as high as 69.9%, and the median progression-free survival time is 12.0 months. It is well comparable with similar drugs and has good safety.

Fluzoparib was approved for the treatment of germline BRCA-mutated (gBRCAm) platinum-sensitive relapsed ovarian cancer in December 2020 and maintenance treatment of platinum-sensitive recurrent ovarian cancer in June 2021. A number of studies on fluzoparib in the field of ovarian cancer are also underway. It is urgent to obtain the real-world data of fluzoparib in the field of ovarian cancer in China. This study will collect information on the baseline characteristics, treatment, and management of ovarian cancer provided in the real world to illustrate the safety and effectiveness of fluzoparib in the treatment of ovarian cancer under the conditions of real clinical practice. It may also include various subgroups of patients with ovarian cancer, which are not involved in the existing phase III registered studies, In order to better understand and explore the use of PARP inhibitors in some patient subgroups and the treatment mode and effect of PARP inhibitors in the treatment of this disease.

ELIGIBILITY:
Inclusion Criteria:

1. Sign informed consent and voluntarily join the study;
2. Epithelial ovarian cancer, fallopian tube cancer, or primary peritoneal cancer diagnosed by histology or cytology;
3. ≥ 18 years old;
4. The investigator determined that the patient could receive fluzoparib monotherapy or combination therapy;
5. For patients with fertility, effective contraceptive methods should be used during the study period and within 90 days after the last administration of fluzoparib

Exclusion Criteria:

1. There is evidence that the patient is a pregnant or lactating woman;
2. Participating in any research with intervention measures other than routine clinical practice; 3. The researcher judges other situations that are not suitable for inclusion in the study;

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with epithelial ovarian cancer, fallopian tube cancer or primary peritoneal cancer had decided to use Fluzoparibb at the time of enrollment in this study
Sampling Method: Non-Probability Sample
Enrollment: 490 (Estimated)
Dates: Start 2022-01-14 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
incidence of ≥ grade 3 Hematology related adverse event according to NCI CTCAE v5.0 | 30 days after the last dose of fluzoparib
  the safety of fluzoparib in ovarian cancer under real-world conditions, especially Incidence of Hematology related adverse reactions ≥ grade 3

SECONDARY OUTCOMES:
incidence of other adverse event according to NCI CTCAE v5.0 | 30 days after the last dose of fluzoparib
  the occasional or rare adverse events of fluzoparib in ovarian cancer under real-world conditions
overall survival (OS) | 6 years
  Overall survival, defined as time from first administration fluzoparib to documented death. To assess clinical effectiveness of fluzoparib monotherapy or combination therapy involved in this study by assessment of overall survival (OS) in patients with Ovarian Cancer. Patients will be followed up once 3-6 months at least
Progression free survival (PFS) | 6 years
  Progression-free survival, defined as time from first administration fluzoparib to documented disease progression or death from any cause after baseline, whichever occurs first;. To assess clinical effectiveness of fluzoparib monotherapy or combination therapy involved in this study by assessment of progression free survival (PFS) in patients with Ovarian Cancer. Patients will be followed up once 3-6 months at least.
Objective Response Rate (ORR) | 6 years
  Objective Response Rate, defined as percentage of patients with complete or partial response according to local assessments. To assess clinical effectiveness of fluzoparib monotherapy or combination therapy involved in this study by assessment of objective response rate (ORR) in patients with Ovarian Cancer. Patients will be followed up once 12 weeks at least.
Disease Control Rate (DCR) | 6 years
  Disease Control Rate, defined as percentage of patients with complete or partial response or stable disease according to local assessments. To assess clinical effectiveness of fluzoparib monotherapy or combination therapy involved in this study by assessment of disease control rate (DCR) in patients with Ovarian Cancer. Patients will be followed up once 12 weeks at least.
Duration Of Therapy（DOT） | 6 years
  Duration Of Therapy, defined as the time from first administration fluzoparib to the permanent cessation of fluzoparib (including death).
Tumor marker expression level | 6 years
  Measurements of tumor biomarkers, such as : CA125, HRD, BRCA, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China